CLINICAL TRIAL: NCT02039713
Title: Evaluation of Effectiveness and Safety of DESyne in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: DESyne in Routine Clinical Practice
Acronym: IRIS DESYNE
Status: Terminated | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Amg Korea Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2014-01
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease
Keywords: DeSyne; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IRIS DeSyne: DeSyne drug eluting stent group
  Interventions: Device: DeSyne drug eluting stent group

INTERVENTIONS:
Device: DeSyne drug eluting stent group

SUMMARY:
The purpose of this study is to evaluate effectiveness and safety of DESyne in Routine Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and more
* Intervention with DeSyne drug eluting coronary stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with DeSyne drug eluting coronary stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with DeSyne stent
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Composite event rate | 1year
  Death, non fatal myocardial infarction, Target Vessel Revascularization

SECONDARY OUTCOMES:
All death | 5year
Cardiac death | 5year
Myocardial infarction | 5year
Composite event of death or myocardial infarction | 5year
Composite event of cardiac death or myocardial infarction | 5year
Target Vessel revascularization | 5year
Target Lesion revascularization | 5year
Stent thrombosis | 5year
  stent thrombosis as classified by an Academic Research Consortium
Stroke | 5year
Procedural success | 3day
  defined as less than 30% residual stenosis at the completion of procedure without death or Q wave myocardial infarction or urgent revascularization
  participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Sam Anyang Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Konkuk University Chungju hospital, Chungju
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Kwangju Christian Hospital, Kwangju
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.